CLINICAL TRIAL: NCT03096054
Title: A Cancer Research UK (CR-UK) Phase I Trial of LY3143921 a Cdc7 Inhibitor in Adult Patients with Advanced Solid Tumours
Brief Title: A CR-UK Phase I Trial of LY3143921
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CRUKD/17/004; 2016-001245-80 (EudraCT Number)
Record Dates: First submitted 2017-03-15; First posted 2017-03-30 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: A. Colorectal Cancer; B. High Grade Serous Ovarian Cancer; C. Non Small-cell Lung Cancer (squamous Cell Variant); D. Squamous Carcinoma of the Oesophagus; E. Squamous Carcinoma of the Head and Neck (HPV Negative); F. Urothelial Cancer; G. Breast Cancer (triple Negative Type); H. Pancreatic Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1 a dose escalation (Experimental): Phase where groups of patients will receive increasing doses of LY3143921 hydrate to find a safe dose and a dose that best targets the cancer cells.
  Interventions: Drug: LY3143921 hydrate
- Part 2 an expansion (Experimental): Phase where a larger group of patients will receive the highest dose of LY3143921 hydrate considered to be safe from Part 1, to find out more about how the drug is working.
  Interventions: Drug: LY3143921 hydrate

INTERVENTIONS:
Drug: LY3143921 hydrate — LY3143921 hydrate will be administered orally on a daily schedule. Each cycle of treatment will consist of 21 days, and patients may initially receive up to 12 cycles. If the patient is benefitting, they may continue beyond 12 cycles.

SUMMARY:
This clinical study is looking at a drug called LY3143921 hydrate (a Cdc7 inhibitor) in adult patients with advanced solid tumours. The main aims are to find out the maximum dose of LY3143921 hydrate that can be given safely to patients, more about the potential side effects and how they can be treated

DETAILED DESCRIPTION:
This clinical study is looking at a drug called LY3143921 hydrate (a Cdc7 inhibitor). Cdc7 helps our cells replicate correctly. In normal cells, Cdc7 is usually found at a low level, but can reach higher levels in cancer cells. This is often the case in certain types of solid tumour cancers, which we will focus on in this study. It is thought that giving LY3143921 hydrate will block the function of Cdc7 and will affect cancer cells by stopping their replication and causing them to die. LY3143921 hydrate looks promising in laboratory studies and studies in animals.

This clinical study has two parts:

Part 1 - a 'dose escalation' phase where groups of patients will receive increasing doses of LY3143921 hydrate to find a safe dose and a dose that best targets the cancer cells. This part of the trial is now closed.

Part 2 - an 'expansion' phase where a larger group of patients will receive the highest dose of LY3143921 hydrate considered to be safe from Part 1, to find out more about how the drug is working.

ELIGIBILITY:
Inclusion Criteria

1. Histologically proven advanced or metastatic solid tumours, refractory to conventional treatment, or for which no conventional therapy exists or is declined by the patient.

   For Phase Ia (dose escalation): Enriched for patients with tumours commonly associated with p53 mutation or loss of function:
   1. Colorectal cancer (CRC)
   2. High grade serous ovarian cancer (HGSOC)
   3. Non small-cell lung cancer (NSCLC, squamous cell variant)
   4. Squamous carcinoma of the oesophagus
   5. Squamous carcinoma of the head and neck (HPV negative)
   6. Urothelial cancer
   7. Breast cancer (triple negative type)
   8. Pancreatic cancer

   For Phase Ib (expansion cohorts): Cohort 1: patients with metastatic CRC; Cohort 2: patients with squamous NSCLC and Cohort 3: patients with solid tumours commonly associated with p53 mutation or loss of function (as described above for the Phase 1a part of the trial).
   * Consent for pre-treatment and post-treatment fresh tumour biopsy samples in a minimum of six patients in expansion Cohorts 1 and 3, optional for all other patients.
   * Consent for pre and post treatment skin punch biopsy
2. Life expectancy of at least 12 weeks.
3. Written (signed and dated) informed consent and be capable of co-operating with treatment and follow-up.
4. World Health Organisation (WHO) performance status of 0 or 1
5. Haematological and biochemical indices within the ranges shown below:

   Laboratory Test Value required
   * Haemoglobin (Hb) ≥ 9.0 g/dL (no prior transfusion) or ≥ 10.0 g/dL (transfusion within last 4 weeks)
   * Absolute neutrophil count ≥1.5 x 10^9/L
   * Platelet count ≥100 x 10^9/L
   * Serum bilirubin ≤1.5 x upper limit of normal (ULN)
   * Alanine amino-transferase (ALT) and aspartate amino-transferase (AST) ≤ 2.5 x (ULN) (or ≤5 x ULN in the presence of liver metastasis)

   Either:
   * Calculated creatinine clearance (using the Wright or C&G formula) > 50 mL/min
   * INR or PTT** ≤1.5 x ULN
   * Albumin ≥ 80% of the lower limit of normal

     * **Therapeutic INR values (2.0-3.0) are acceptable to confirm eligibility for patients who are taking concomitant warfarin
6. Age 18 years or over.
7. Consent must be given for use of archived tumour samples for all patients.
8. Disease must be either evaluable or measurable using RECIST v1.1 criteria.

Exclusion Criteria:

1. Systemic anti-cancer therapy (with the exception of life-long hormone suppression such as luteinising hormone-releasing hormone (LHRH) agents in prostate cancer) or another investigational agent during the previous 4 weeks (6 weeks for nitrosureas, Mitomycin-C) is not permitted. Previous use of radiotherapy is permitted except where there has been a large volume of bone marrow irradiated or where the irradiated lesion is the only one suitable for RECIST measurability.
2. Ongoing toxic manifestations of previous treatments (Grade 2 or greater according to NCI-CTCAE v4.02) with the exception of alopecia or certain Grade 2 toxicities, which in the opinion of the investigator and Sponsor should not exclude the patient - these should be discussed on a case by case basis.
3. Symptomatic brain metastases or spinal cord compression.
4. Significant baseline hypotension (<90mmgHg systolic or <50 mmHg diastolic).
5. Uncontrolled hypertension (>160mmHg/100mmHg).
6. Patients with a known left ventricular ejection fraction (LVEF) <50%. An echocardiogram (ECHO) must be performed in all patients.
7. Women of child-bearing potential3 (or are already pregnant or lactating). However, those patients who meet the following points are considered eligible:

   * Have a negative serum or urine pregnancy test before enrolment and;
   * Agree to use two forms of contraception (one effective form plus a barrier method) [oral, injected or implanted hormonal contraception and condom; intra-uterine device and condom; diaphragm with spermicidal gel and condom] or agree to sexual abstinence4, effective from the first administration of LY3143921 hydrate, throughout the trial and for six months afterwards.
8. Male patients with partners of child-bearing potential. However, those patients who meet the following points are considered eligible:

   * Agree to take measures not to father children by using a barrier method of contraception [condom plus spermicide] or to sexual abstinence4 effective from the first administration of LY3143921 hydrate, throughout the trial and for six months afterwards.
   * Men with partners of child-bearing potential must also be willing to ensure that their partner uses an effective method of contraception for the same duration for example, hormonal contraception, intra-uterine device, diaphragm with spermicidal gel or sexual abstinence.
   * Men with pregnant or lactating partners must be advised to use barrier method contraception (for example, condom plus spermicidal gel) to prevent exposure of the foetus or neonate.
9. No major surgery within 4 weeks prior to the patient receiving Cycle 1 Day-7 (for dose escalation) or C1 Day1 (for dose expansion). If minor surgery has been performed within 2 weeks of the start of trial treatment then patients must have recovered, and the sponsor and CI should be notified of the nature of this and agree to patient inclusion.
10. At high medical risk because of non-malignant systemic disease including active uncontrolled infection.
11. Known to be serologically positive for Hepatitis B, Hepatitis C or Human Immunodeficiency Virus (HIV) (mandatory testing not required).
12. Significant cardiovascular disease as defined by:

    1. History of congestive heart failure requiring therapy
    2. History of unstable angina pectoris or myocardial infarction up to 6 months prior to trial entry
    3. Presence of severe valvular heart disease
    4. Presence of a ventricular arrhythmia requiring treatment
13. Past history of corneal ulceration, dry eye syndrome, glaucoma. Contact lenses should also be avoided during participation in the trial.
14. Any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.
15. Is a participant or plans to participate in another interventional clinical trial, whilst taking part in this Phase I study of LY3143921 hydrate. Participation in an observational trial or interventional clinical trial which does not involve administration of an IMP and which would not place an unacceptable burden on the patient in the opinion of the Investigator and Medical Advisor would be acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Determination of the maximal dose | 28 days including the single dose on Cycle 1 Day-7
  Determining the maximal dose at which no more than one patient out of up to six patients at the same dose level experience a highly probably or probably drug related DLT and determining the schedule of administration at which the MTD is established.
  Determining causality of each AE to LY3143921 hydrate and grading severity according to NCI -CTCAE Version 4.02.

SECONDARY OUTCOMES:
Determine the Cmax | Up to 21 time points from first dose
  LY3143921 hydrate levels will be measured in serum by liquid chromatography mass spectrometry (LCMS) according to agreed standard operating procedures (SOPs) and validated methods.
Determine the Tmax | Up to 21 time points from first dose
  LY3143921 hydrate levels will be measured in serum by liquid chromatography mass spectrometry (LCMS) according to agreed standard operating procedures (SOPs) and validated methods.
Determine the area under the curve (AUC) | Up to 21 time points from first dose
  LY3143921 hydrate levels will be measured in serum by liquid chromatography mass spectrometry (LCMS) according to agreed standard operating procedures (SOPs) and validated methods.
Determine the plasma halflife, | Up to 21 time points from first dose
  LY3143921 hydrate levels will be measured in serum by liquid chromatography mass spectrometry (LCMS) according to agreed standard operating procedures (SOPs) and validated methods.
Determine the volume of distribution | Up to 21 time points from first dose
  LY3143921 hydrate levels will be measured in serum by liquid chromatography mass spectrometry (LCMS) according to agreed standard operating procedures (SOPs) and validated methods.
Determine the clearance of LY3143921 hydrate | Up to 21 time points from first dose
  LY3143921 hydrate levels will be measured in serum by liquid chromatography mass spectrometry (LCMS) according to agreed standard operating procedures (SOPs) and validated methods.
Determine the response rate | Database lock- 4 weeks after the last patient last
  Free survival rate of patients treated with LY3143921 hydrate according to the Response
Determine the median progression | Database lock- 4 weeks after the last patient last
  Free survival rate of patients treated with LY3143921 hydrate according to the Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - Cancer Centre, Belfast City Hospital, Belfast
  - Western General Hospital, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Northern Centre for Cancer Care, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No